CLINICAL TRIAL: NCT01181180
Title: The Effect of Fluids Consumption in the Elderly on Balance and Gait Function - A Single Blind Randomized Control Trial
Brief Title: The Effect of Fluids Consumption on Balance and Gait Function in Old Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SOR496510CTIL; SORMBS4965 (Other Grant/Funding Number: Goldman fundation)
Record Dates: First submitted 2010-05-27; First posted 2010-08-13 (Estimated); Last update posted 2024-04-19 (Actual); Status verified 2010-07

CONDITIONS: Aging; Dehydration
Keywords: Ageing; Balance control; Falls; dehydration
MeSH Terms: conditions — Dehydration | interventions — Drinking; Aging

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- water consumation treatment (Experimental)
  Interventions: Dietary Supplement: water consumption
- no water consumption treatment (Placebo Comparator)
  Interventions: Dietary Supplement: water consumption

INTERVENTIONS:
Dietary Supplement: water consumption — The effect of water consumption on postural stability of old adults (65 years old and over) will be measured using RCT study design
  Other Names: balance in older adults

SUMMARY:
Experimental design overview The proposed project is a prospective experimental RCT study design. Independent old adults(age 65 years old and older) who do not suffer from balance problems willing to participate in the study will be tested before and after water consumption to explore whether there are differences in balance control as a result of dehydration.

DETAILED DESCRIPTION:
Experimental design overview The proposed project is a prospective experimental study design. independent old adults(age 65 years old and older) who do not suffer from balance problems willing to participate in the study will be tested with well-established measuring techniques of Balance control before and 2 hours after mineral water consumption (1 liter) in the movement and Rehabilitation Laboratory at BGU. An automated algorithm will be used to extract standardized stabilogram-diffusion parameters from each of the COP data sets collected during quiet standing. These parameters include diffusion coefficients, critical displacement, critical time and scaling exponents for both lateral and anterior-posterior sway directions (Collins & De Luca, 1993). For each of the conditions (before and 1 hour after the use of Ritalin) in three task conditions single task; dual task (concentrating and identifying specific music); and just Listening to a relaxing music. Participants will be required to stand on the platform 10 times for 30 s. For each trial, they will be instructed to sway as little as possible.

ELIGIBILITY:
Inclusion Criteria:

* age 65 years old and older
* independent elderly adults
* do not suffer from balance problems
* mini-mental score 24 and above

Exclusion Criteria:

* old adults who suffer from neurological disease or stroke
* old adults who suffer from psychiatric state
* old adults who suffer from orthopedic condition (1/2 a year after a fracture in the lower limb)
* old adults who suffer from heart conditions
* old adults who suffer from blindness

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Postural sway measures | Time 1: pre test' and hour later time 2: post testinng proceedure

CONTACTS AND LOCATIONS:
Overall Officials: Melzer Itshak, PhD, Principal Investigator — Ben-gurion University of the Negev, Beer-Sheva, Israel; Bar-David Yair, MD, Study Director — Soroka University Medical Centar; Snir Yorm, MD, Study Chair — Soroka University Medical Center
Locations (1):
- SorokaUMC, Beersheba, Israel